CLINICAL TRIAL: NCT00918632
Title: A Phase I Open-Label Study In Healthy Volunteers To Compare The Plasma Pharmacokinetics of Polymorph Form XLI AG-013736 In The Fasted And Fed State
Brief Title: Food Effect Study Of AG-013736 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A4061053
Record Dates: First submitted 2009-06-08; First posted 2009-06-11 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Healthy Volunteers
Keywords: food-effect pharmacokinetics AG-013736 food fasting
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (ABC) (Other): The following treatments will be administered in the following order A -> B-> C
  1. Treatment A = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered after overnight fasting
  2. Treatment B = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a high-fat, high-calorie meal.
  3. Treatment C = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a moderate-fat, standard-calorie meal.
  Interventions: Drug: AG-013736
- Sequence 2 (ACB) (Other): The following treatments will be administered in the following order A -> C -> B
  1. Treatment A = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered after overnight fasting
  2. Treatment B = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a high-fat, high-calorie meal.
  3. Treatment C = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a moderate-fat, standard-calorie meal.
  Interventions: Drug: AG-013736
- Sequence 3 (BCA) (Other): The following treatments will be administered in the following order B -> C -> A
  1. Treatment A = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered after overnight fasting
  2. Treatment B = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a high-fat, high-calorie meal.
  3. Treatment C = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a moderate-fat, standard-calorie meal.
  Interventions: Drug: AG-013736
- Sequence 4 (BAC) (Other): The following treatments will be administered in the following order B -> A -> C
  1. Treatment A = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered after overnight fasting
  2. Treatment B = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a high-fat, high-calorie meal.
  3. Treatment C = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a moderate-fat, standard-calorie meal.
  Interventions: Drug: AG-013736
- Sequence 5 (CAB) (Other): The following treatments will be administered in the following order C -> A -> B
  1. Treatment A = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered after overnight fasting
  2. Treatment B = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a high-fat, high-calorie meal.
  3. Treatment C = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a moderate-fat, standard-calorie meal.
  Interventions: Drug: AG-013736
- Sequence 6 (CBA) (Other): The following treatments will be administered in the following order C -> B -> A
  1. Treatment A = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered after overnight fasting
  2. Treatment B = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a high-fat, high-calorie meal.
  3. Treatment C = AG-013736 polymorph Form XLI film-coated immediate release (FCIR) tablet administered with a moderate-fat, standard-calorie meal.
  Interventions: Drug: AG-013736

INTERVENTIONS:
Drug: AG-013736 — A single dose of a FCIR tablet of AG-013736 will be administered under overnight fasting (Treatment A), high-fat, high-calorie meal (Treatment B), or moderate-fat, standard-calorie meal (Treatment C) in the following order A -> B -> C. Each of these treatments will be separated by a 7 day washout period.
  Arms: Sequence 1 (ABC)
Drug: AG-013736 — A single dose of a FCIR tablet of AG-013736 will be administered under overnight fasting (Treatment A), high-fat, high-calorie meal (Treatment B), or moderate-fat, standard-calorie meal (Treatment C) in the following order A -> C -> B. Each of these treatments will be separated by a 7 day washout period.
  Arms: Sequence 2 (ACB)
Drug: AG-013736 — A single dose of an FCIR tablet of AG-013736 will be administered under overnight fasting (Treatment A), high-fat, high-calorie meal (Treatment B), or moderate-fat, standard-calorie meal (Treatment C) in the following order B -> C -> A. Each of these treatments will be separated by a 7 day washout period.
  Arms: Sequence 3 (BCA)
Drug: AG-013736 — A single dose of a FCIR tablet of AG-013736 will be administered under overnight fasting (Treatment A), high-fat, high-calorie meal (Treatment B), or moderate-fat, standard-calorie meal (Treatment C) in the following order B -> A -> C. Each of these treatments will be separated by a 7 day washout period.
  Arms: Sequence 4 (BAC)
Drug: AG-013736 — A single dose of a FCIR tablet of AG-013736 will be administered under overnight fasting (Treatment A), high-fat, high-calorie meal (Treatment B), or moderate-fat, standard-calorie meal (Treatment C) in the following order C -> A -> B. Each of these treatments will be separated by a 7 day washout period.
  Arms: Sequence 5 (CAB)
Drug: AG-013736 — A single dose of a FCIR tablet of AG-013736 will be administered under overnight fasting (Treatment A), high-fat, high-calorie meal (Treatment B), or moderate-fat, standard-calorie meal (Treatment C) in the following order C -> B -> A. Each of these treatments will be separated by a 7 day washout period.
  Arms: Sequence 6 (CBA)

SUMMARY:
The study is designed to evaluate the effect of food on typical blood levels obtained after oral dosing of AG-013736. Drug levels in blood will be compared after an overnight fast and a high-fat, high-calorie meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead Electrocardiogram (ECG) and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.

Exclusion Criteria:

* Evidence of history of clinically significant blood, kidney, endocrine, gastrointestinal, heart, liver, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* Active smokers or users of other tobacco products as well as users of certain drugs.
* Pregnant or nursing females; females of childbearing potential, including those with tubal ligation. To be considered for enrollment, women of 45 to 55 years of age who are postmenopausal (defined as being amenorrheic for at least 2 years) must have confirmatory Follicle-stimulating hormone (FSH) test results at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To assess the effect of a high-fat, high-calorie meal and overnight fasting on polymorph Form XLI AG-013736 plasma pharmacokinetics following a single 5 mg oral dose in healthy volunteers. | 2 months

SECONDARY OUTCOMES:
To assess the effect of a moderate-fat, standardized meal and overnight fasting on polymorph Form XLI AG-013736 plasma pharmacokinetics following a single 5 mg oral dose in healthy volunteers. | 2 months
To assess the safety and tolerability of single-dose polymorph Form XLI AG-013736 when administered with a high-fat, high-calorie meal, a moderate-fat, standard-calorie meal and overnight fasting in healthy volunteers. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061053&StudyName=Food%20Effect%20Study%20Of%20AG-013736%20In%20Healthy%20Volunteers